CLINICAL TRIAL: NCT06775132
Title: Associations Between Dietary Intake and Cardiometabolic and Gut Microbiota Outcomes in Singapore Adults
Brief Title: Associations Between Dietary Intake and Cardiometabolic and Gut Microbiota Outcomes
Status: Recruiting | Type: Observational
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant Professor, National University of Singapore
Other Study IDs: S27
Record Dates: First submitted 2025-01-01; First posted 2025-01-14 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cardiometabolic Risk Factors; Gut -Microbiota; Skin Condition; Cognitive Ability, General; Sleep Quality
Keywords: Endothelial progenitor cells; Gut microbiota; Cardiovascular diseases risk factors; MoCA; Advanced glycation end products
MeSH Terms: conditions — Skin Diseases; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — plasma, serum, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Younger population: Age 21-64
- Middle-aged and older population: Age 65-80

SUMMARY:
This cross-sectional study aims to investigate the associations between dietary intake, cardiometabolic health markers, and gut microbiota composition in Singapore adults.

DETAILED DESCRIPTION:
Diet plays a crucial role in maintaining overall health, and changes in dietary patterns are increasingly recognized as major contributors to chronic disease development. Inadequate dietary intake and poor diet quality have been linked to increased risks of cardiometabolic diseases and disruptions in gut microbiota composition. However, most studies investigating these associations have been conducted on Western populations, and there is a lack of research focusing on Asian populations. Given the genetic, metabolic, and dietary differences between Western and Asian populations, examining these associations in an Asian population is essential for a deeper understanding of population-specific risk factors and health outcomes. Therefore, there is an urgent need to assess the associations between dietary intake, cardiometabolic health, and gut microbiota composition in Asian population.

This cross-sectional study aims to investigate the associations between dietary intake, cardiometabolic health markers, and gut microbiota composition in Singapore adults.

Findings from this study will offer valuable insights into the relationship between diet, cardiometabolic health, and the gut microbiota in this population. In addition, this research may identify specific dietary patterns or nutrients that offer greater benefit for cardiometabolic and gut health. In turn, these findings can contribute to the improvement of current dietary guidelines aimed at promoting better cardiometabolic and gut microbiota outcomes for the broader Singaporean population.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give informed consent
2. Adults 21-80 years old
3. English-literate
4. Have venous access sufficient to allow for blood sampling as per the protocol
5. No drastic change of diet for the past 1 year
6. If taking medication, has been consistently taking antihypertensive/cholesterol-lowering/type-2 diabetic medication for more than 5 years prior to starting the study.

Exclusion Criteria:

1. Taking dietary supplements and fermented foods, which may impact the gut microbiota (e.g. antibiotics, prebiotics, probiotics, yogurt, kimchi) 2 months before starting the 1st study visit only.
2. Taking dietary supplements or medications, which may impact sleep outcomes (e.g. Nutritional Shakes (e.g. Ensure), tryptophan, 5-hydroxytryptophan or melatonin supplementations) 1 month before starting the study.
3. Taking dietary supplements which may impact the eye outcomes (e.g. Vitamin A, vitamin A-containing multivitamin) 2 months before starting the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Singapore adults
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Dietary intake | Day 7
  Use a 3-day food record to document dietary intake
Blood pressure | Day 1
  Systolic and diastolic blood pressure (in mmHg) will be measured by a blood pressure monitor.
Blood lipid lipoprotein profile | Day 1
  Total cholesterol, LDL, HDL, and triglyceride concentration in the blood will be measured
Fasting blood glucose | Day 1
  Glucose concentration in the blood will be measured
Endothelial Progenitor Cell Count | Day 1
  Endothelial functions are determined by the percentage of endothelial progenitor cells (CD34+/KDR+) expression in peripheral blood mononuclear cells
Fecal short chain fatty acid (SCFA) concentration | Day 1
  SCFA concentration in the blood will be measured
Trimethylamine N-oxide (TMAO) | Day 1
  Trimethylamine N-oxide (TMAO) concentration in the blood will be measured
Fecal bile acids | Day 1
  Bile acids concentration will be determined from fecal samples of the subjects
Fecal zonulin | Day 1
  Zonulin concentration will be determined from fecal samples of the subjects
Fecal calprotectin | Day 1
  Calprotectin concentration will be determined from fecal samples of the subjects
Estimated Glomerular Filtration Rate (eGFR) | Day 1
  The estimated Glomerular Filtration Rate (eGFR) of the subjects will be measured from the blood

SECONDARY OUTCOMES:
Sleep quality-Pittsburgh Sleep Quality Index Questionnaire | Day 1
  Pittsburgh Sleep Quality Index Questionnaire (PSQI) will be used to assess the sleep quality. Overall score ranging from 0 to 21 points, where lower scores denote a healthier sleep quality.
Cognitive function | Day 1
  Use Montreal Cognitive Assessment (MoCA) questionnaires to assess cognitive function. A score of 26 or above (out of 30) is generally considered normal, though adjustments may be made for educational level.
Skin carotenoid concentration | Day 1
  Skin carotenoid concentration: This can be measured by Resonance Raman Spectroscopy, the unit is skin carotenoid score, a higher score means optimal, lower score means poor condition of skin carotenoids.
Macular Pigment Optical Density (MPOD) | Day 1
  Macular Pigment Optical Density (MPOD): A measurement of macular pigment of the eye using a heterochromatic flicker photometry device. The measurements are in arbitrary units.
The Global Physical Activity Questionnaire (GPAQ) | Day 1
  The Global Physical Activity Questionnaire (GPAQ) will be used to assess physical activity levels in three areas: work, transport, and leisure. It measures activity in terms of frequency, duration, and intensity, generating a score in metabolic equivalents (METs). Higher MET values indicate higher levels of physical activity.
The Perceived Stress Scale (PSS-10) | Day 1
  The Perceived Stress Scale (PSS-10) will be used to assess the level of perceived stress over the past month. The scale consists of 10 items scored on a 5-point Likert scale (0 = never to 4 = very often), with a total score ranging from 0 to 40. Higher scores indicate greater perceived stress.
The Beck Anxiety Inventory (BAI) | Day 1
  The Beck Anxiety Inventory (BAI) will be used to measure the severity of anxiety symptoms. It consists of 21 questions scored on a 4-point Likert scale (0 = not at all to 3 = severely). The total score ranges from 0 to 63, with higher scores reflecting more severe anxiety symptoms.
The Beck Depression Inventory-II (BDI-II) | Day 1
  The Beck Depression Inventory-II (BDI-II) will be used to assess the severity of depressive symptoms over the past two weeks. It contains 21 questions scored on a 4-point scale (0 = no symptoms to 3 = severe symptoms). Total scores range from 0 to 63, with higher scores indicating more severe depression.
Visual acuity | Day 1
  Participants will read out letters on a ETDRS LogMAR chart at a fixed distance where letters becomes smaller as it goes down the chart. Tests results will be recorded in number of letters read, where the more letters the better the outcome.
Visual function questionnaire 25 | Day 1
  A questionnaire to for participants to self-evaluate their perception of their current eye health based on general vision, ocular pain, near activities, distance activities, vision specific functions, driving, color vision and peripheral vision. The best possible score is 100 and worst possible score is 0.
Skin advanced glycation end products (AGE) levels | Day 1
  Skin advanced glycation end products (AGE) levels: Measurement of skin advanced glycation end products level using a skin autofluorescence device, where participants wlll be instructed to place their forearm over the device and a light will be shone and a reading can be captured by detecting fluorescence. The results will be presented as arbitrary units.

OTHER OUTCOMES:
Anthopometric measurements | Day 1
  Height, weight, and waist circumference will be measured for each subject

CONTACTS AND LOCATIONS:
Overall Officials: Jung Eun Kim, Principal Investigator — Department of Food Science and Technology, National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No